CLINICAL TRIAL: NCT07333677
Title: A Safety and Efficacy Study of in Vivo CAR-T (HN2301) for Refractory Graves' Disease
Brief Title: In Vivo CAR-T for Refractory Graves' Disease
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2025-805
Record Dates: First submitted 2025-12-20; First posted 2026-01-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-11

CONDITIONS: Graves' Disease
Keywords: refractory Graves' disease; TSH receptor antibody; in vivo CAR-T
MeSH Terms: conditions — Graves Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- In Vivo CAR-T Therapy for Refractory Graves' Disease (Experimental): Participants with refractory Graves' disease will receive three to five intraveneous administrations of In Vivo CAR-T (HN2301).
  Interventions: Biological: In Vivo CAR-T Therapy

INTERVENTIONS:
Biological: In Vivo CAR-T Therapy — Participants will receive 3 to 5 intravenous administrations of HN2301, given once every 2 days, according to the study dosing regimen.
  Other Names: HN2301

SUMMARY:
Graves' disease is an autoimmune thyroid disorder characterized by the production of autoantibodies against the thyroid-stimulating hormone receptor (TRAb), leading to excessive thyroid hormone secretion and systemic manifestations. A subset of patients develop refractory disease, failing to achieve durable remission despite prolonged antithyroid therapy.

This study aims to evaluate the safety and efficacy of HN2301, an in vivo CAR-T therapy in which host T lymphocytes are engineered and transformed to functional CAR-T cells via CD8 antibody-coated LNP delivery of CD19 CAR-mRNA. Participants with refractory Graves' disease will receive three to five administrations of HN2301 and will be regularly monitored for changes in thyroid function, TRAb levels, clinical response, and treatment-related adverse events. The study will provide preliminary evidence on whether HN2301 can induce sustained remission of refractory Graves' disease.

ELIGIBILITY:
Inclusion Criteria (Participants must meet all of the following criteria to be eligible for this study):

* Age 18-75 years (inclusive), male or female.
* Refractory Graves' disease, defined as meeting at least one of the following: a) Continuous antithyroid drug (ATD) therapy for ≥3 years without achieving criteria for ATD discontinuation; b) Meeting criteria for ATD discontinuation but experiencing ≥2 relapses after ATD withdrawal.
* Positive serum TRAb.
* Willing to use effective contraception for 12 months after study drug administration.
* Voluntarily agrees to participate in the study, has signed the informed consent form, and is able to comply with study procedures and follow-up requirements.

Exclusion Criteria (Participants meeting any of the following criteria will be excluded from the study):

* History of severe drug allergy or known allergic predisposition.
* Presence or suspected presence of uncontrolled active infection.
* History of major organ transplantation (e.g., heart, lung, liver, kidney) or bone marrow/hematopoietic stem cell transplantation.
* Presence of significant heart disease, such as angina, myocardial infarction, heart failure, or clinically significant arrhythmias.
* Receipt of any mRNA-LNP product or other lipid nanoparticle (LNP)-based therapy within the past 2 years.
* Receipt of a live vaccine within 30 days prior to screening.
* History of malignant tumors.
* Positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb) with peripheral blood HBV DNA above the detection limit; positive hepatitis C virus (HCV) antibody with detectable HCV RNA; positive human immunodeficiency virus (HIV) antibody; or positive syphilis test.
* Presence of psychiatric disorders or severe cognitive impairment.
* Hematologic dysfuction at screening, defined as any of the following: a. Neutrophil count < 1.8 × 10⁹/L, b. Hemoglobin < 110 g/L, c. Platelet count < 50 × 10⁹/L
* Impaired liver function, defined as any of the following: Alanine aminotransferase (ALT) > 3 × ULN, Aspartate aminotransferase (AST) > 3 × ULN, Total bilirubin > 2.5 × ULN.
* Impaired renal function: creatinine clearance rate (CrCl) < 60 mL/min (Cockcroft-Gault formula).
* Left ventricular ejection fraction (LVEF) < 55%.
* Coagulation abnormalities, defined as either: International normalized ratio (INR) > 1.5 × ULN, Prothrombin time (PT) > 1.5 × ULN
* Pregnant or breastfeeding women.
* Any other condition that, in the opinion of the investigator, would make the participant unsuitable for the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of Adverse Events (AEs) | From baseline to 3 months after infusion of HN2301
  Assessment of the incidence and severity of treatment-emergent adverse events (AEs) occurring within 3 months after drug administration at the recommended dose.
Remission of Graves' disease | From baseline to 12 months after infusion of HN2301
  Proportion of remission will be calculated throughout 12 months after initial dose of HN2301. Remission is defined as euthyroid status without anti-thyroid medication.

SECONDARY OUTCOMES:
Proportion of participants with ≥50% reduction of anti-thyrotropin receptor antibody (TRAb) | From baseline to 12 months after infusion of HN2301
  Percentage of participants achieving a ≥50% reduction of TRAb throughout 12 months after initial dose of HN2301, as compared with baseline.
Proportion of participants with ≥50% reduction of thyroid stimulating immunoglobulin (TSI) | From baseline to 12 months after infusion of HN2301
  Percentage of participants achieving a ≥50% reduction of TSI througout 12 months after initial dose of HN2301, as compared with baseline.
Change of TRAb levels compared to baseline | From baseline to 12 months after infusion of HN2301
  TRAb levels will be measured from baseline to 12 months after initial dose of HN2301
Change of TSI levels compared to baseline | From baseline to 12 months after infusion of HN2301
  TSI levels will be measured from baseline to 12 months after initial dose of HN2301
Change of thyroid gland volume compared to baseline | From baseline to 12 months after infusion of HN2301
  Size of thyroid will be measured and calculated by ultrasound from baseline to 12 months after initial dose of HN2301
Change of thyroid peroxidase antibody (TPOAb) levels compared to baseline | From baseline to 12 months after infusion of HN2301
  TPOAb levels will be measured from baseline to 12 months after initial dose of HN2301
Change of Thyroglobulin antibody (TgAb) levels compared to baseline | From baseline to 12 months after infusion of HN2301
  TgAb levels will be measured from baseline to 12 months after initial dose of HN2301
Proportion of CAR-T cells generated in peripheral blood after HN2301 administration | Day 0 to Day 14
  Proportion of CAR-T cells generated in peripheral blood after infusion of HN2301
Time to peak CAR-T Cell generation in peripheral blood after HN2301 administration | Day 0 to Day 14
  Time to reach the peak level of CAR-T cells generated in peripheral blood after infusion of HN2301
Dynamic change of CAR gene copy number in peripheral blood after HN2301 administration | Day 0 to Day 14
Dynamic change of peripheral blood B lymphocyte cell count after HN2301 administration | From baseline to 12 months after infusion of HN2301
Dynamic change of serum interleukin-6 after HN2301 administration | From baseline to 12 months after infusion of HN2301
Dynamic change of serum tumor necrosis factor α (TNF-α) after HN2301 administration | From baseline to 12 months after infusion of HN2301
Dynamic change of serum immunoglobulin levels after HN2301 administration | From baseline to 12 months after infusion of HN2301

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: After publication.
Access Criteria: IPD and supporting information will be avaible to researchers upon reasonable request (e.g. with a practical and meaningful research proposal).